#### INSTITUTE BOARD DECISION

MEETING DATE: 28.09.2023

MEETING TIME: 14:00

MEETING NUMBER: 2023/33

DECISION NUMBER: 2023/33-69

The Department of Obstetrics and Gynecology Nursing at our institute has decided to accept the thesis suggestion of Ümmü Gülsüm COŞKUN, a student in the Obstetrics and Gynecology Nursing Master's Program, with the title stated below:

**Thesis Title:** "Evaluation of the Efficacy of Manual Pressure and Local Cold Spray Application in Reducing Pain from Human Anti-D Immunoglobulin Injection in Pregnant Women: A Randomized Controlled Study"

## **Supervisor**

Assoc Prof. Dilek Coşkuner Potur

#### **VOLUNTARY CONSENT FORM**

#### Dear Participant;

The research titled "Evaluation of the Efficacy of Manual Pressure and Local Cold Spray Application in Reducing Pain Caused by Human Anti-D Immunoglobulin Injection in Pregnant Women: A Randomized Controlled Study" was planned by ümmü Gülsüm Coşkun under the supervision of Assoc. Prof. Dr. Dilek Coskuner POTUR. The purpose of this research is to determine the effect of manual pressure and local cold spray application in reducing the pain caused by Human Anti-D Immunoglobulin injection. The research is planned to be conducted with 129 pregnant women. You will be administered the prescribed Anti-D Immunoglobulin injection as part of the study. Before the application, the Introductory Information Form, Fear of Pain Scale III, and after the application of local cold spray, an injection will be administered, followed by the Visual Comparison Scale and Injection Satisfaction Scale. Filling out these forms will take approximately 5-10 minutes. During the research, the confidentiality of your information will be prioritized, and the information you provide will be used only for scientific research purposes. Voluntariness is the basis for participating in this study. At any stage of the study, you can voluntarily withdraw with or without providing reasons. The financial obligation of the study belongs to the researchers, and no payment or fee will be requested from voluntary participants. You will only be asked to fill out the forms and scales used in the research. For our research to yield accurate results, it is important to answer all items in the surveys correctly. Thank you for your participation.

Dear participant, you have the right to refuse to participate in the research. With notice, you can withdraw from the study at any time or be excluded from the study if deemed necessary by the researcher. If you decline to participate in the research or are removed from the study for any reason, it will not affect your work life. You will not incur any financial responsibility for the expenses related to the research, and no payment will be made to you. All information obtained from you will be kept confidential and used only in the mentioned research.

Contributions to Science and Medicine: Due to the widespread use of injection applications and the experience of pain associated with it, many studies are being conducted to reduce injection pain. The Human Anti-D Immunoglobulin injection, which is both original and common, easily prevents complications that may arise due to possible blood incompatibility. Therefore, in order to minimize the pain intensity of sensitive groups such as pregnant women, low-cost, effective, and reliable methods should be used in the clinical setting. Our research aims to demonstrate the effectiveness of manual pressure and local cold spray application, promote their widespread use in the clinical setting, and increase the injection satisfaction of pregnant women. Thus, pregnant women will be able to complete the existing treatment for potential complications due to blood incompatibility with minimal pain from injections in an easy and effective manner.

DATE .../.../2023

VOLUNTARY CONSENT FORM (LOCAL COLD SPRAY APPLICATION GROUP)

I have read all the explanations in the Informed Consent Form. I have been provided with

written and verbal explanations about the research described above, its subject, and purpose by

the researchers Ümmü Gülsüm Coşkun under the supervision of Assoc. Prof. Dr. Dilek

Coşkuner POTUR. After receiving this information, I was invited to participate in such research

as a "participant." I know that I can voluntarily participate in the research and withdraw from

the research at any time with or without reasons. I believe that great care and respect will be

shown to the confidentiality of my information during this research. I trust that my personal

information will be carefully protected during the use of research results for scientific purposes.

I agree to participate in this research voluntarily, without any pressure or coercion.

Participant's Name - Surname: Signature:

Researcher's Name - Surname: Signature:

DATE .../.../2023

VOLUNTARY CONSENT FORM (MANUAL PRESSURE APPLICATION GROUP)

I have read all the explanations in the Informed Consent Form. I have been provided with

written and verbal explanations about the research described above, its subject, and purpose by

the researchers Ümmü Gülsüm Coşkun under the supervision of Assoc. Prof. Dr. Dilek

Coşkuner POTUR. After receiving this information, I was invited to participate in such research

as a "participant." I know that I can voluntarily participate in the research and withdraw from

the research at any time with or without reasons. I believe that great care and respect will be

shown to the confidentiality of my information during this research. I trust that my personal

information will be carefully protected during the use of research results for scientific purposes.

I agree to participate in this research voluntarily, without any pressure or coercion.

Participant's Name - Surname: Signature:

Researcher's Name - Surname: Signature:

DATE .../.../2023

VOLUNTARY CONSENT FORM (CONTROL GROUP)

I have read all the explanations in the Informed Consent Form. I have been provided with

written and verbal explanations about the research described above, its subject, and purpose by

the researchers Ümmü Gülsüm Coşkun under the supervision of Assoc. Prof. Dr. Dilek

Coşkuner POTUR. After receiving this information, I was invited to participate in such research

as a "participant." I know that I can voluntarily participate in the research and withdraw from

the research at any time with or without reasons. I believe that great care and respect will be

shown to the confidentiality of my information during this research. I trust that my personal

information will be carefully protected during the use of research results for scientific purposes.

I agree to participate in this research voluntarily, without any pressure or coercion.

Participant's Name - Surname: Signature:

Researcher's Name - Surname: Signature:

#### INTRODUCTORY INFORMATION FORM

This study is designed to determine the impact of manual pressure and local cold spray application on reducing the pain of Human Anti-D Immunoglobulin injection. Your responses are crucial for the reliability of the research. Therefore, it is highly important that you assess honestly and meticulously in a way that reflects you, to achieve scientific results. We appreciate your participation in this research.

| Age: | | | |
|---|---|---|---|
| Height: | | | |
| Weight: | | | |
| BMI: | | | |
| Employment Status : a) Yes b) No | | | |
| Education Level: a) Primary School | l b) High School c) Univer | sity | |
| Job : | | | |
| Blood Type: | | | |
| | Gravida :<br>Miscarriage: | | Parite : |
| vious Use of Human Immunoglobulin | Anti-D Injection: a) Yes | b) No | |
| Hemodynamic Parameters | | | |
| od Pressure:<br>se:<br>piratory Rate: | After Injection Blood Presssure: Pulse: Respiratory Rate: Oxygen Saturation: | | |
| | Job: Blood Type: Obstetric Parameters t Menstual Period: ivery Type: | Height: Weight: BMI: Employment Status: a) Yes b) No Education Level: a) Primary School b) High School c) Univer Job: Blood Type: Obstetric Parameters t Menstual Period: Gravida: Miscarriage: vious Use of Human Immunoglobulin Anti-D Injection: a) Yes Hemodynamic Parameters ore Injection After Injection od Pressure: Blood Presssure: se: Pulse: repiratory Rate: Respiratory Rate: | Height: Weight: BMI: Employment Status : a) Yes b) No Education Level : a) Primary School b) High School c) University Job : Blood Type: Obstetric Parameters t Menstual Period: Gravida : ivery Type: Miscarriage: vious Use of Human Immunoglobulin Anti-D Injection: a) Yes b) No Hemodynamic Parameters ore Injection After Injection od Pressure: Blood Presssure: se: Pulse: Respiratory Rate: |

# VISUAL ANALOG SCALE



# INJECTION SATISFACTION SCALE



### FEAR OF PAIN QUESTIONNAIRE – III

| Name: | Date: |
|-------|-------|

INSTRUCTIONS: The items listed below describe painful experiences. Please look at each item and think about how FEARFUL you are of experiencing the PAIN associated with each item. If you have never experienced the PAIN of a particular item, please answer on the basis of how FEARFUL you expect you would be if you had such an experience. Circle one number for each item below to rate your FEAR OF PAIN in relation to each event.

| an experience. Circle one number for each item below to face your FEAR OF FAIN in relation to each event. | | | | | | |
|---|---|---|---|---|---|---|
| | | Not<br>At All | A Little | A Fair<br>Amount | Very<br>Much | Extreme |
| I FEAR the PAIN associated with: | | | | | | |
| 1. | Being in an automobile accident. | 1 | 2 | 3 | 4 | 5 |
| 2. | Biting your tongue while eating. | 1 | 2 | 3 | 4 | 5 |
| 3. | Breaking your arm. | 1 | 2 | 3 | 4 | 5 |
| 4. | Cutting your tongue licking an envelope. | 1 | 2 | 3 | 4 | 5 |
| 5. | Having a heavy object hit you in the head. | 1 | 2 | 3 | 4 | 5 |
| 6. | Breaking your leg. | 1 | 2 | 3 | 4 | 5 |
| 7. | Hitting a sensitive bone in your elbow – your "funny bone." | 1 | 2 | 3 | 4 | 5 |
| 8. | Having a blood sample drawn with a hypodermic needle. | 1 | 2 | 3 | 4 | 5 |
| 9. | Having someone slam a heavy car door on your hand. | 1 | 2 | 3 | 4 | 5 |
| 10. | Falling down a flight of concrete stairs. | 1 | 2 | 3 | 4 | 5 |
| 11. | Receiving an injection in your arm. | 1 | 2 | 3 | 4 | 5 |
| 12. | Burning your fingers with a match. | 1 | 2 | 3 | 4 | 5 |
| 13. | Breaking your neck. | 1 | 2 | 3 | 4 | 5 |
| 14. | Receiving an injection in your hip/buttocks. | 1 | 2 | 3 | 4 | 5 |
| 15. | Having a deep splinter in the sole of your foot probed and removed with tweezers. | 1 | 2 | 3 | 4 | 5 |
| 16. | Having an eye doctor remove a foreign particle stuck in your eye. | 1 | 2 | 3 | 4 | 5 |
| 17. | Receiving an injection in your mouth. | 1 | 2 | 3 | 4 | 5 |
| 18. | Being burned on your face by a lit cigarette. | 1 | 2 | 3 | 4 | 5 |
| 19. | Getting a paper-cut on your finger. | 1 | 2 | 3 | 4 | 5 |
| 20. | Receiving stitches in your lip. | 1 | 2 | 3 | 4 | 5 |
| 21. | Having a foot doctor remove a wart from your foot with a sharp instrument. | 1 | 2 | 3 | 4 | 5 |
| 22. | Cutting yourself while shaving with a sharp razor. | 1 | 2 | 3 | 4 | 5 |
| 23. | Gulping a hot drink before it has cooled. | 1 | 2 | 3 | 4 | 5 |
| 24. | Getting strong soap in both your eyes while bathing or showering. | 1 | 2 | 3 | 4 | 5 |
| 25. | Having a terminal illness that causes you daily pain. | 1 | 2 | 3 | 4 | 5 |
| 26. | Having a tooth pulled. | 1 | 2 | 3 | 4 | 5 |
| 27. | Vomiting repeatedly because of food poisoning. | 1 | 2 | 3 | 4 | 5 |
| 28. | Having sand or dust blow into your eyes. | 1 | 2 | 3 | 4 | 5 |
| 29. | Having one of your teeth drilled. | 1 | 2 | 3 | 4 | 5 |
| 30. | Having a muscle cramp. | 1 | 2 | 3 | 4 | 5 |